CLINICAL TRIAL: NCT00005497
Title: Risk Factors for Pulmonary Hypertension of the Newborn
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5015; R01HL058763 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-10

CONDITIONS: Persistent Fetal Circulation Syndrome; Lung Diseases
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome; Lung Diseases

SUMMARY:
To conduct a multicenter case-control study of persistent pulmonary hypertension of the newborn (PPHN) in relation to maternal exposure to smoking and non-steroidal anti-inflammatory drugs (NSAIDs). Also, to assess other potential antenatal risk factors and collect and store buccal cell specimens for future analyses.

DETAILED DESCRIPTION:
BACKGROUND:

Persistent pulmonary hypertension of the newborn (PPHN), previously called persistent fetal circulation, is a birth defect affecting approximately 1 in 1250 liveborn term infants; even with complex and high-risk interventions, PPHN results in substantial mortality and morbidity. This defect results from the inappropriate muscularization of fetal pulmonary vessels, and experimental and human evidence consistently suggests that maternal cigarette smoking and antenatal exposure to NSAIDs, particularly aspirin or ibuprofen, may play a role in the etiology of this condition. Because these exposures are quite prevalent (e.g., ibuprofen is currently taken in the first trimester or later in pregnancy by 15 percent and 3.2 percent of women, respectively), testing these hypotheses is of considerable public health importance.

DESIGN NARRATIVE:

The multicenter study had a case-control design. There were 560 case infants with PPHN and four controls per case (2240). All controls were drawn from the birth hospitals of cases; half the controls had malformations other than PPHN, and half had normal formations. Cases and controls were identified within five months of birth at 88 birth and tertiary hospitals in the areas surrounding Boston, Philadelphia, and Toronto. Mothers of subjects were interviewed by telephone within six months of delivery; a standardized questionnaire inquired in detail about demographic factors; reproductive, medical, and pregnancy illness histories; medication use (including a detailed focus on use of over-the-counter analgesic/antipyretic medications), smoking, and nutrition. Because of emerging genetic research suggesting an effect of NSAIDs on pathways possibly related to the etiology of PPHN, buccal swabs were also collected and stored for future analyses. Exposure prevalences were compared between mothers of cases and controls and relative risks were estimated, controlling for potential confounding factors.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-04; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allen Mitchell — Boston University

REFERENCES:
- [Background] Hernandez-Diaz S, Werler MM, Walker AM, Mitchell AA. Folic acid antagonists during pregnancy and the risk of birth defects. N Engl J Med. 2000 Nov 30;343(22):1608-14. doi: 10.1056/NEJM200011303432204. PMID 11096168
- [Background] Hernandez-Diaz S, Werler MM, Louik C, Mitchell AA. Risk of gestational hypertension in relation to folic acid supplementation during pregnancy. Am J Epidemiol. 2002 Nov 1;156(9):806-12. doi: 10.1093/aje/kwf129. PMID 12396998
- [Background] Louik C, Werler MM, Mitchell AA. Erythromycin use during pregnancy in relation to pyloric stenosis. Am J Obstet Gynecol. 2002 Feb;186(2):288-90. doi: 10.1067/mob.2002.119718. PMID 11854652
- [Background] Hernan MA, Hernandez-Diaz S, Werler MM, Mitchell AA. Causal knowledge as a prerequisite for confounding evaluation: an application to birth defects epidemiology. Am J Epidemiol. 2002 Jan 15;155(2):176-84. doi: 10.1093/aje/155.2.176. PMID 11790682
- [Background] Hernandez-Diaz S, Werler MM, Walker AM, Mitchell AA. Neural tube defects in relation to use of folic acid antagonists during pregnancy. Am J Epidemiol. 2001 May 15;153(10):961-8. doi: 10.1093/aje/153.10.961. PMID 11384952
- [Background] Waller DK, Tita AT, Werler MM, Mitchell AA. Association between prepregnancy maternal body mass index and the risk of having an infant with a congenital diaphragmatic hernia. Birth Defects Res A Clin Mol Teratol. 2003 Jan;67(1):73-6. doi: 10.1002/bdra.10003. PMID 12749387
- [Background] Werler MM, Louik C, Mitchell AA. Epidemiologic analysis of maternal factors and amniotic band defects. Birth Defects Res A Clin Mol Teratol. 2003 Jan;67(1):68-72. doi: 10.1002/bdra.10001. PMID 12749386
- [Background] Hernandez-Diaz S, Hernan MA, Meyer K, Werler MM, Mitchell AA. Case-crossover and case-time-control designs in birth defects epidemiology. Am J Epidemiol. 2003 Aug 15;158(4):385-91. doi: 10.1093/aje/kwg144. PMID 12915504
- [Background] de Jong-Van den Berg LT, Hernandez-Diaz S, Werler MM, Louik C, Mitchell AA. Trends and predictors of folic acid awareness and periconceptional use in pregnant women. Am J Obstet Gynecol. 2005 Jan;192(1):121-8. doi: 10.1016/j.ajog.2004.05.085. PMID 15672013
- [Background] Hernandez-Diaz S, Wu XF, Hayes C, Werler MM, Ashok TD, Badovinac R, Kelsey KT, Mitchell AA. Methylenetetrahydrofolate reductase polymorphisms and the risk of gestational hypertension. Epidemiology. 2005 Sep;16(5):628-34. doi: 10.1097/01.ede.0000172132.13513.e0. PMID 16135938